CLINICAL TRIAL: NCT00959127
Title: A Study of ARRY-438162 (MEK162) in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-162-111
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumors; Advanced or Metastatic Biliary Cancer; Metastatic Colorectal Cancer
Keywords: Colorectal Adenocarcinoma; Colon Cancer; Rectal Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARRY-438162 (MEK 162) (Experimental)
  Interventions: Drug: ARRY-438162 (MEK162), MEK inhibitor; oral

INTERVENTIONS:
Drug: ARRY-438162 (MEK162), MEK inhibitor; oral — Part 1: multiple dose, escalating; Part 2: multiple dose, single schedule; Part 3: multiple dose, single schedule.

SUMMARY:
This is a Phase 1 study during which patients with advanced solid tumors will receive investigational study drug ARRY-438162 (MEK162).

This study has 3 parts. In the first part, patients with advanced solid tumors will receive increasing doses of study drug in order to achieve the highest dose of the study drug possible that will not cause unacceptable side effects. Approximately 30 patients from the US will be enrolled in Part 1. (Active, not recruiting)

In the second part of the study, patients with advanced or metastatic biliary cancer will receive the best dose of study drug determined from the first part of the study and will be followed to see what side effects and effectiveness the study drug has, if any, in treating the cancer. Approximately 25 patients from the US will be enrolled in Part 2. (Active, not recruiting)

In the third part of the study, patients with metastatic colorectal cancer (CRC) will receive the best dose of the study drug determined from the first part of the study and will be followed to see what side effects and effectiveness the study drug has, if any, in treating the cancer. Approximately 25 patients with KRAS mutation (Active, not recruiting) and 15 patients with BRAF mutation (Active, not recruiting) from the US will be enrolled in Part 3.

ELIGIBILITY:
Key Inclusion Criteria (for Part 3):

* A histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma which is metastatic (measurable disease).
* Documented KRAS- or BRAF- tumor mutation.
* Previously treated with or unsuitable for treatment with 5-Fluorouracil (5-FU), oxaliplatin, irinotecan and, if available, bevacizumab.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Additional criteria exist.

Key Exclusion Criteria (for Part 3):

* Uncontrolled or symptomatic brain metastases (if the patient has brain metastases and is on steroids, the steroid dose must have been stable for at least 30 days).
* History of central serous retinopathy, retinopathy visible at baseline that would be considered a risk factor for central serous retinopathy or retinal vein occlusion.
* Concomitant malignancies or previous malignancies with less than a 2-year disease free interval at the time of enrollment; patients with adequately resected basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or stage A low grade prostate cancer may enroll irrespective of the time of diagnosis.
* Prior treatment with a MEK inhibitor.
* Treatment with prior chemotherapy, anticancer immunotherapy, monoclonal antibodies or other protein or peptide therapeutics within 21 days of the first dose of study drug.
* Treatment with a small molecule targeted agent or anticancer hormonal therapy within 14 days of the first dose of study drug.
* Treatment with prior radiotherapy within 28 days of initiating study drug (if the radiation portal covered ≤ 10% of the bone marrow reserve, the patient may be enrolled irrespective of the end date of radiotherapy).
* Major surgery within 4 weeks or minor surgery within 7 days prior to the first dose of study drug.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis C, and/or active hepatitis B.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of the study drug. | Part 1, one year
Characterize the safety profile of the study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | Parts 1, 2 and 3: two years
Characterize the pharmacokinetics (PK) of the study drug and metabolite. | Parts 1, 2 and 3: two years

SECONDARY OUTCOMES:
Assess the efficacy of the study drug in terms of tumor response, duration of response, duration of stable disease, progression-free survival and overall survival. | Parts 1, 2 and 3: two years
Assess possible PK/pharmacodynamic (PD) or PK/efficacy and safety correlations. | Parts 1, 2 and 3: two years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas